CLINICAL TRIAL: NCT06644170
Title: A Phase 1 Study of a Second Psilocybin Group Retreat for Partial Responders With Anxiety Associated With Metastatic Cancer
Brief Title: A Second Psilocybin Group Therapy for the Treatment of Cancer-Related Anxiety in Partial Responders With Metastatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Steven & Alexandra Cohen Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1124860; NCI-2024-08058 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20619 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2024-10-11; First posted 2024-10-16 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Metastatic Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Behavior Therapy; Psychotherapy, Group; Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (psilocybin, group therapy) (Experimental): Patients receive psilocybin PO with optional booster dose on day 0. Patients attend an individual prep visit on day -1 and an individual integration visit on day 1. Patients also attend group preparation visits on days -14, -7 and -1 and group integration visits on days 1, 8, 22 and 36.
  Interventions: Behavioral: Behavioral Intervention; Behavioral: Group Therapy; Drug: Psilocybin; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Behavioral Intervention — Attend individual visits
  Other Names: Psychedelic therapy
Behavioral: Group Therapy — Attend group visits
Drug: Psilocybin — Given PO
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase I trial tests the safety and side effects of a second episode of psilocybin-assisted group therapy and how well it works in treating anxiety and distress in patients with cancer that has spread from where it first started (primary site) to other places in the body (metastatic) and had a partial response to their first retreat. Up to 50% of patients with metastatic cancer have clinically significant anxiety and unaddressed anxiety and distress may add to the suffering caused by cancer itself. Psilocybin, a psychedelic drug, is made using an extract from the psilocybe mushroom, also known as "magic mushrooms". Psilocybin binds to serotonin receptors (natural body chemicals that control moods) on brain cells producing intense changes in mood, including anxiety. This may change perceptions and patterns of thinking in ways that may decrease anxiety. Group therapy may reduce stress and improve the well-being and quality of life of patients with metastatic cancer. A second episode of psilocybin-assisted group therapy may be safe, tolerable and or effective in treating anxiety and distress in partial responders with metastatic cancer.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive psilocybin orally (PO) with optional booster dose on day 0. Patients attend an individual prep visit on day -1 and an individual integration visit on day 1. Patients also attend group preparation visits on days -14, -7 and -1 and group integration visits on days 1, 8, 22 and 36.

After completion of study treatment, patients are followed up at 2, 3, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Participation in BACK002, with outcome measures that showed: a low Mystical Experience Questionnaire (MEQ) score, OR a small (or negative) Hospital Anxiety and Depression Scale (HADS) change score, OR a last HADS score that was 11 or greater, OR who have experienced a recurrence in their symptoms of anxiety or depression since completing the 6 month follow-up
* A diagnosis of metastatic solid tumor, or incurable hematologic malignancy that has been accepted by a physician in a medical record
* Measurable disease is not required
* Previous treatment with chemotherapy: There are no minimum or maximum prior lines of chemotherapy
* 18-85 years of age
* Required performance status, including the appropriate scale. Eastern Cooperative Oncology Group (ECOG) 0-2
* Hematocrit > 20
* Platelets (Plt) > 20K
* Liver function tests 1.5 x normal
* Creatinine 1.5 x normal
* Subjects of childbearing potential must be willing to use an effective contraceptive method from study enrollment until at least 1 month after receiving the investigational agent(s)
* Must be at least 4 weeks after surgery or radiotherapy at study entry, but can be receiving oral or intravenous (IV) chemotherapy if those schedules can be adjusted around the medication session date
* Motivated to participate in a group study and able in the research team's judgment to participate in the small group effectively
* On pre-enrollment screening tests, they will have clinically significant anxiety or depressive symptoms as defined by a score of 11 or greater on the HADS-Total
* English speaking - able to understand the process of consent and the risk and benefits associated with the study, and able to give written informed consent. This is a pilot study, and if future larger studies are designed, consideration will be given for non-english-speaking subjects
* Must be willing to sign a medical release for the investigators to communicate directly with their treating clinicians (mental health professional or oncologist) and doctors to confirm a medication and/or medical history
* Must provide at least one adult who is in contact with the participant at least once a day when the participant is at home for the first day after returning home who is able to verbally monitor participant-reported changes in the behavior and able to notify research staff of behavior changes that may require research staff assessment
* (In BACK002, participants were required to taper off selective serotonin reuptake inhibitors [SSRIs] in this study they will be allowed to continue.) Must provide a review of any SSRI use since completing BACK002
* Must avoid taking any psychiatric medications or starting a new psychiatric medication during the study. Should participant's doctor recommend starting a new psychiatric medication, participant will be required to notify the study team and the subject would withdraw from the study. (Use of as needed [prn] benzodiazepines is allowed but high dose chronic benzodiazepine use must be reviewed by the principal investigator [PI]. Use of prn gabapentoids is allowed but high dose chronic gabapentoid use must be reviewed by the PI.)
* Must provide a contact (relative, spouse, close friend, or other caregiver) who is willing and able to be reached by the research team in the event that the participant becomes suicidal
* If the potential participant is of childbearing potential, they must have a negative pregnancy test at baseline and prior to the medication dosing session, and must agree to use adequate birth control
* Are willing to commit to preparation sessions, medication dosing sessions, integration sessions, to complete evaluation instruments and commit to be contacted for all necessary telephone contacts
* Must have had serum lab tests within 1 week of the retreat showing values for potassium (K), magnesium (Mg), and calcium in the normal range. (Electrolyte repletion and rechecking of serum labs is allowed to establish eligibility.)

Exclusion Criteria:

* Brain metastases that have not been treated
* Uncontrolled or concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnancy, breastfeeding, or expecting to conceive or father children for the duration of the trial through 30 days after receipt of investigational agent(s)
* Personal or immediate family history of schizophrenia, bipolar affective disorder, delusion disorder, paranoid disorder, or schizoaffective disorder
* Suicidal ideation with a Columbia-Suicidality Severity Rating Scale (C-SSRS) ≥ 3
* Current substance abuse disorder (although prospective subjects will not be excluded for reasonable alcohol use that does not meet criteria for alcohol use disorder or marijuana use that does not meet criteria for substance use disorder)
* Unstable neurological or medical condition; history of seizure, chronic/severe headaches
* Any use of psychedelic drugs in high doses (psilocybin > 2 grams of dried mushrooms, lysergic acid diethylamide (LSD) > 200 micrograms) within the prior 3 months (microdosing will not require exclusion but participants would have to agree to discontinue microdosing 1 month before study entry)
* Use of tramadol, due to the potential for serotonin syndrome with concomitant use of psilocybin
* Individuals who are on MAOI (monoamine oxidase inhibitors) or who have a known sensitivity to the drug or its metabolites. Psilocybin is contraindicated in medications that are known UGT (UDP-glucuronosyltransferase) enzyme modulators
* Baseline prolongation of QT/corrected QT (QTc) interval (e.g., demonstration on an eligibility 12-lead electrocardiogram [ECG] of a QTc interval > 450 milliseconds [ms])
* A history of additional risk factors for Torsade de Points (including but not limited to: heart failure, hypokalemia, family history of long QT syndrome)
* The use of concomitant medications that prolong the QT/QTc interval
* Any history of cardiovascular disease such as history of myocardial infarction or congestive heart failure or cardiac arrhythmia
* Concomitant use of efavirenz (an antiviral) which cannot be tapered
* Concomitant use of serotonin-acting supplements due to their potential for interaction with psilocybin, including oxitriptan (5-HTP), St John's Wort, and 'brain food' supplements

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-11-19 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | At time of first exposure up to the date of the last questionnaire at 24 weeks
  AEs will be defined as any untoward medical occurrence in a clinical investigation subject administered a medicinal product. AEs will be graded in severity using mild, moderate and severe. Occurrence of any adverse event graded severe on the Common Terminology Criteria for Adverse Events patient-reported questionnaires. Descriptive statistics will be used to analyze all adverse events, and in particular severe adverse events.

SECONDARY OUTCOMES:
Change in anxiety and depression | At day -14 up to day 28
  Changes will be measured using the Hospital Anxiety and Depression Scale. For each group size, the "effect size" of change will be estimated, where effect size is defined as the mean change divided by the standard deviation of change. Assessment of anxiety and depression will be descriptive.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony L. Back, MD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-01-28): https://cdn.clinicaltrials.gov/large-docs/70/NCT06644170/ICF_000.pdf